CLINICAL TRIAL: NCT04310995
Title: Effect of Nicorandil, Diltiazem or Isosorbide Mononitrate for Oral Antispastic Therapy After Coronary Artery Bypass Grafting Using Radial Artery Grafts - a Pilot Randomized Controlled Trial
Brief Title: Different Anti-Spastic Therapy Strategies After CABG Using Radial Artery Grafts
Acronym: ASRAB-Pilot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Chugai Pharma China (Unknown)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Vice President of RuijinHospital, Professor and Director, Department of Cardiac Surgery, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIG-IIS001C
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Bypass Graft; Radial Artery Grafts; Antispastic Therapy; Pilot Study
Keywords: CABG; Radial artery grafts; Antispastic; Nicorandil; Diltiazem; Isosorbide Mononitrate
MeSH Terms: interventions — Nicorandil; Diltiazem; isosorbide-5-mononitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nicorandil (Experimental)
  Interventions: Drug: Nicorandil 5mg tid
- Diltiazem (Experimental)
  Interventions: Drug: Diltiazem 180mg qd
- Isosorbide Mononitrate (Experimental)
  Interventions: Drug: Isosorbide Mononitrate 50mg qd

INTERVENTIONS:
Drug: Nicorandil 5mg tid — oral Nicorandil Tablets 5mg (5mg per tablet) three times daily for 24 weeks
  Arms: Nicorandil
Drug: Diltiazem 180mg qd — oral Diltiazem Sustained-release Tables180mg (90 mg per tablet) once daily for 24 weeks
  Arms: Diltiazem
Drug: Isosorbide Mononitrate 50mg qd — oral Isosorbide Mononitrate Sustained-release Capsules 50 mg (50mg per capsule) once daily for 24 weeks
  Arms: Isosorbide Mononitrate

SUMMARY:
The Pilot study will be a single-center, randomized, open-label, active-controlled trial. After CABG surgery using Radial Artery Grafts (RA-CABG) and signing the informed consent, all patients will be screened according to the inclusion and exclusion criteria. Estimated 150 patients will be enrolled and randomized by ratio 1:1:1 to receive either Nicorandil (5mg tid po) or Diltiazem (180mg qd po) or Isosorbide Mononitrate (50mg qd po). Follow-up visits will be conducted at Week 1, 4, 12, and 24 after surgery. The last evaluation of study endpoints and other adverse events will be at Week 24.

The pilot study is designed to explore the angiography outcomes of grafts and cardiovascular outcomes of patients, as well as safety outcomes among different anti-spastic regimens after RA-CABG.

DETAILED DESCRIPTION:
After having signed informed consent (Day 1-3), eligible subjects who have successfully received first RA-CABG surgery (Day 0) will be screened for enrollment. All subjects (150 patients) will be randomized in a 1:1:1 ratio into 3 groups. Group A will receive oral Nicorandil (5mg tid) monotherapy; Group B will receive oral Diltiazem (180mg qd) monotherapy; and Group C will receive Isosorbide Mononitrate (50mg qd) monotherapy. Three groups will continue intervention treatment for 24 weeks after RA-CABG surgery. All subjects will receive follow-up visits (clinic visit or phone visit) at Week 1, 4, 12, and 24 after surgery.

All subjects will receive first CCTA (or CAG) to evaluate the graft outcome at Week 1 and second CCTA (or CAG) to evaluate the graft outcome at Week 24 after RA-CABG surgery. And all subjects will be evaluated angina relief based on the Canadian Cardiovascular Society (CCS) angina grading and the Seattle Angina Questionnaire. And the time to first major adverse cardiovascular event (MACE), which include all-cause mortality, myocardial infarction, stroke and unplanned revascularization, will be collected. And other safety outcomes will be evaluated, including the rate of hypotension, the proportion of concomitant medications with ACEI/ARB/ARNI drugs and proportion of SAEs and concerned AEs.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old，
* Male or female patients，
* Have signed informed consent，
* Have successfully received a RA-CABG surgery 1-3 days ago.

Exclusion Criteria:

* Previously experienced an allergy to active ingredients and/or excipients of experimental drugs,
* Hypotension (defined as systolic blood pressure < 90mmHg or diastolic blood pressure < 60mmHg) after surgery,
* Acute myocardial infarction, pulmonary congestion or cardiogenic shock after surgery,
* Concomitant medications with phosphodiesterase-5 inhibitors such as sildenafil, vardenafil, tadalafil, etc,
* Pathological sinus node syndrome, degree II or III atrioventricular block without cardiac pacemaker,
* With contraindications for coronary computed tomography angiography (CCTA) or coronary arteriography (CAG) examination, such as iodine allergy, etc. note: patients with renal insufficiency or even end-stage receiving hemodialysis but can be tolerated by CCTA or CAG examination (judged by investigators) are eligible for inclusion,
* History or evidence of ongoing alcohol or drug abuse,
* Life expectancy < 1 year judged by investigators,
* Other inappropriate situations judged by investigators .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
the rate of RA graft failure at Week 1 | at Week 1
  CCTA or CAG will be used to evaluate the RA graft outcome at Week 1 after RA-CABG. The definition of RA-graft outcomes will refer to the modified Fitzgibbon classification criteria. When RA-graft outcome conform to the Grade B, O or S, the result will be judged as the graft failure.
the rate of RA graft failure at Week 24 | at Week 24
  CCTA or CAG will be used to evaluate the RA graft outcome at at Week 24 after RA-CABG. The definition of RA-graft outcomes will refer to the modified Fitzgibbon classification criteria. When RA-graft outcome conform to the Grade B, O or S, the result will be judged as the graft failure.

SECONDARY OUTCOMES:
the time to first Major Adverse Cardiovascular Events (MACE) | within 24 weeks
  MACE will include all-cause death, myocardial infarction, stroke and unplanned revascularization.
the proportion of subjects with angina recurrence | within 24 weeks
  The angina symptoms will be evaluated by Canadian Cardiovascular Society angina grade and Seattle Angina Questionnaires.
the proportion of subjects with at least one hypotension occurrence | within 24 weeks
  Subjects' blood pressure will be measured by sitting in the clinic or by using a sphygmomanometer outside the hospital (recorded on the diary card). Systolic blood pressure < 90mmHg or diastolic blood pressure < 60mmHg will be recorded as "hypotension" as defined in the study.
the proportion of subjects with ACEI/ARB/ARNI withdrawal | within 24 weeks
  The subjects who stop using ACEI/ARB/ARNI ≥20% of the time during the study period will be recorded as "ACEI/ARB/ARNI withdrawal" as defined in the study.
the proportion of subjects with serious adverse events (SAEs) and concerned adverse events (AEs) | within 24 weeks
  SAE will include death; life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability/incapacity; a congenital anomaly/birth defect in the offspring of the patient; judged to be medically significant (including laboratory abnormalities). concerned AEs will include: cardiac arrest, reoperation, incision complications, pulmonary infection, respiratory failure, new atrial fibrillation/atrial flutter, permanent pacemaker implantation, and gastrointestinal hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD.PhD, Principal Investigator — Ruijin Hospital; Yunpeng Zhu, MD, Study Director — Ruijin Hospital; Mario FL Gaudino, MD, Principal Investigator — Weill Cornell Medicine NewYork Presbyterian Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, China

REFERENCES:
- [Derived] Zhu Y, Zhang W, Qin K, Liu Y, Yao H, Wang Z, Ye X, Zhou M, Li H, Qiu J, Xu H, Sun Y, Gaudino M, Zhao Q. Effects of Nicorandil, Isosorbide Mononitrate, or Diltiazem on Radial Artery Grafts After CABG: The Randomized ASRAB-Pilot Trial. Circ Cardiovasc Interv. 2025 Apr;18(4):e014542. doi: 10.1161/CIRCINTERVENTIONS.124.014542. Epub 2025 Mar 24. PMID 40123490